CLINICAL TRIAL: NCT03888859
Title: Phase 1, Open-label, Three Routes IV, Intratumoral Injections and Intra-hepatic Artery Dose-escalation Clinical Study to Evaluate the Safety and Efficacy of ET1402L1-ARTEMIS™2™ T- Cells in AFP Expressing Hepatocellular Carcinoma (HCC)
Brief Title: ET1402L1-ARTEMIS™2 T Cells in Alpha Fetoprotein (AFP) Expressing Hepatocellular Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Eureka Therapeutics Inc. (Industry); Aeon Therapeutics (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2017LSL-C002
Record Dates: First submitted 2019-02-01; First posted 2019-03-25 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Liver Neoplasms; Metastatic Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous (i.v.) arm (Experimental): autologous ET1402L1-ARTEMIS™2 T cells administered by intravenous (IV) infusion
  Interventions: Biological: ET1402L1-ARTEMIS™ T cells -IV
- Intra-hepatic artery (i.a.) arm (Experimental): autologous ET1402L1-ARTEMIS™2 T cells administered by intra-hepatic artery (IA) infusion
  Interventions: Biological: ET1402L1-ARTEMIS™ T cells -intra-hepatic artery
- Intratumoral Injections (i.t.) arm (Experimental): autologous ET1402L1-ARTEMIS™2 T cells administered by intratumoral injections (i.t.) infusion
  Interventions: Biological: ET1402L1-ARTEMIS™ T cells -Intratumoral Injections

INTERVENTIONS:
Biological: ET1402L1-ARTEMIS™ T cells -IV — Autologous T cells transduced with lentivirus encoding an anti-AFP (ET1402L1) -ARTEMIS™2 expression construct -intravenous (i.v.) arm
  Arms: Intravenous (i.v.) arm
Biological: ET1402L1-ARTEMIS™ T cells -intra-hepatic artery — Autologous T cells transduced with lentivirus encoding an anti-AFP (ET1402L1) -ARTEMIS™2 expression construct: intra-hepatic artery (i.a.) arm
  Arms: Intra-hepatic artery (i.a.) arm
Biological: ET1402L1-ARTEMIS™ T cells -Intratumoral Injections — Autologous T cells transduced with lentivirus encoding an anti-AFP (ET1402L1) -ARTEMIS™2 expression construct: Intratumoral Injections (i.t.) arm
  Arms: Intratumoral Injections (i.t.) arm

SUMMARY:
Clinical study to evaluate safety (primary objectives) and efficacy (secondary objective) of ET1402L1-ARTEMIS™2 T cells in patients with alpha fetoprotein positive (AFP+ ) hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The molecular target for ET1402L1-ARTEMIS™2 is human leukocyte antigen (HLA) -A02 complexed with a HLA-A02-restricted peptide of alpha fetoprotein (AFP), which is expressed on 60-80 percent of hepatocellular carcinoma (HCC). ARTEMIS™2 is a second generation ARTEMIS™ receptor engineered with a human antibody domain against the anti-HLA-A02/AFP complex. This clinical study evaluates the safety and pharmacokinetics of ET1402L1-ARTEMIS™2 T-cells in patients with HCC who have no available curative therapeutic options and a poor overall prognosis.

Patients with lesion(s) localized in liver will be enrolled in the intra-hepatic artery (IA) arm or Intratumoral Injections arm, with the ET1402L1-ARTEMIS™2 T-cells administered via intrahepatic artery catheter. Patients with extrahepatic metastasis will be enrolled in the intravenous (IV) arm, with the ET1402L1-ARTEMIS™2 T-cells administered through intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* AFP-expressing HCC and serum AFP >100 ng/mL.
* Abandon or failure in first or second line treatment
* Molecular HLA class I typing confirms participant carries at least one HLA-A02 allele
* Child-Pugh score of A or B, Barcelona Clinic Liver Cancer stage of C or D
* Life expectancy > 4 months
* Karnofsky score ≥70%
* Adequate organ function as defined below:

  1. Patients must have a serum Total bilirubin ≤2 x Upper Limit of Normal (ULN), Alanine transaminase (ALT) and Aspartate transaminase (AST) ≤5 times the institutional ULN.
  2. A pretreatment measured creatinine clearance (absolute value) of ≥ 50 ml/minute
  3. Ejection fraction measured by echocardiogram or Multiple gated acquisition scanning (MUGA) >45% (evaluation done with 6 weeks of screening does not need to be repeated)
  4. Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) or Forced Expiratory Volume in the first second (FEV1)>45% predicted
  5. Absolute neutrophil count (ANC) ≥ 1500/mm3 (10^9/L)
  6. Platelet count ≥ 50,000/mm3 (10^9/L)
* Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients with decompensated cirrhosis: Child-Pugh Score C
* Patients with tumor infiltration in the portal vein, hepatic veins or inferior vena cava that completely blocks circulation in liver.
* Patients with an organ transplantation history
* Patients with dependence on corticosteroids
* Patients with active autoimmune diseases requiring systemic immunosuppressive therapy
* Patients who are currently receiving or received within past 30 days anti-cancer therapy, local treatments for liver tumors (radiotherapy, embolism, ablation) or liver surgery
* Patients currently receiving other investigational treatments (biotherapy, chemotherapy, or radiotherapy)
* Participants with other active malignancies (except non-melanoma skin cancer and cervical cancer) within two years. Patients with a history of successfully-treated tumors with no sign of recurrence in the last two years may be enrolled.
* Patients with other uncontrolled diseases, such as active infections
* Acute or chronic active hepatitis B or hepatitis C.
* Women who are pregnant or breast-feed
* HIV-infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity | 28 days up to 2 years
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the ET1402L1-ARTEMIS™2 T-cells, which is irreversible, or life threatening or CTCAE Grade 3-5. Assessed at all visits.
Frequency of ARTEMIS T cell treatment-related adverse events | Time Frame: 28 days up to 2 years
  Include but not limited to: Fever, chills, nausea, vomiting, jaundice and other gastrointestinal symptoms; Fatigue, hypotension, respiratory distress; Tumor lysis syndrome; Cytokine release syndrome; Neutropenia, thrombocytopenia; Liver and kidney dysfunction. Assessed at all visits.

SECONDARY OUTCOMES:
Rate of disease response by RECIST in the liver | 2 years
  Response rates will be estimated as the percent of patients with objective response (OR)，which was defined as any of complete remission (CR), partial response (PR) at 2 years.
Rate of disease response by RECIST at non-liver sites | 2 years
  Response rates will be estimated as the percent of patients with objective response (OR)，which was defined as any of complete remission (CR), partial response (PR) at 2 years.
Progression free survival (PFS) | at 4 months, 1 year, 2 years
  Progression free survival (PFS) at 4 months, 1 year and 2 years
Median Survival（MS） | at 4 months, 1 year, 2 years
  Median Survival（MS）at 4 months, 1 year and 2 years
Overall survival（OS） | at 2 years
  overall survival（OS）at 2 years
AFP serum levels | 2 years
  Percent change compared to the baseline
Number of ET1402L1-ARTEMIS™2 T cells in peripheral blood | 2 years
  Number of ET1402L1-ARTEMIS™2 T cells in peripheral blood will be presented as Time to peak, Time to baseline level
% of ET1402L1-ARTEMIS™2 T cells in peripheral blood | 2 years
  %of ET1402L1-ARTEMIS™2 T cells in peripheral blood will be presented as Time to peak, Time to baseline level
AFP expression in tumors | 4-8 weeks
  Percent of AFP-positive cells in randomly selected fields in tumor biopsies.
Tmax of serum Interleukin (IL)-2, IL-4, IL-6, IL-10, Tumor necrosis factor(TNF)-α and Interferon gamma (INFγ) | 24 weeks
  Increase or decreases in the amount of serum IL-2, IL-4, IL-6, IL-10, TNF-α and INF-γ produced compared to baseline at time points measured up to 24 weeks since dosing. Data will be presented as time to peak level for Tmax.
AUC of serum IL-2, IL-4, IL-6, IL-10, TNF-α and INFγ | 24 weeks
  Increase or decreases in the amount of serum IL-2, IL-4, IL-6, IL-10, TNF-α and INFγ produced compared to baseline at time points measured up to 24 weeks since dosing. Data will be presented as time to peak level for area under curve (AUC).
Time to baseline for serum IL-2, IL-4, IL-6, IL-10, TNF-α and INFγ | 24 weeks
  Increase or decreases in the amount of IL-2, IL-4, IL-6, IL-10, TNF-α and INFγ produced compared to baseline at time points measured up to 24 weeks since dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Liu, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China